CLINICAL TRIAL: NCT02037997
Title: Chemotherapy in Combination With Erlotinib, or Sequential Chemotherapy for Erlotinib for Treatment, EGFR - TKI Resistance of EGFR Mutations in Patients With NSCLC Randomized Controlled Phase II Clinical Study
Brief Title: Safety and Effectiveness Study of Chemotherapy in Combination With Erlotinib,or Sequential Erlotinib for Treatment in Patients With NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, attending, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CJH-Erlotinib-2013
Record Dates: First submitted 2014-01-02; First posted 2014-01-16 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Non Small Cell Lung Cancer
Keywords: PFS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Pemetrexed; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combination with Erlotinib (Experimental): Erlotinib 150mg qd combination with docetaxel 75mg/m2 or pemetrexed 500mg/m2
  Interventions: Drug: docetaxel; Drug: pemetrexed; Drug: Erlotinib
- sequential chemotherapy for Erlotinib (Active Comparator): docetaxel 75mg/m2 or pemetrexed 500mg/m2，after PD，Erlotinib 150mg qd
  Interventions: Drug: docetaxel; Drug: pemetrexed; Drug: Erlotinib

INTERVENTIONS:
Drug: docetaxel — docetaxel 75mg/m2 ivgtt D1
Drug: pemetrexed — pemetrexed 500mg/m2 ivgtt D1
Drug: Erlotinib — Erlotinib 150mg qd

SUMMARY:
The purpose of this study is to evaluate and compare safety and effectiveness of Chemotherapy in Combination With Erlotinib,or Sequential Erlotinib for Treatment in Patients With EGFR - TKI Resistance of EGFR Mutations

DETAILED DESCRIPTION:
from the first cycle of treatment (day one) to two month after the last cycle

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent
2. ≥18 years
3. According to RECIST 1.1 standard, at least one measurable lesions
4. Histology and cytology confirmed with unfavorable surgical locally advanced stage (stage IIIB) or metastatic NSCLC (IV), Sensitive EGFR gene mutation
5. Palliative treatment has received two medicine first-line platinum-based chemotherapy and EGFR - TKI second-line treatment and objective clinical benefit (CR, PR or SD is more than 6 months), RESIST standard curative effect evaluation for progress
6. PS=0,1,2
7. No serious blood, heart, lung, liver and kidney dysfunction, and immune deficiency
8. Hb≥9g/dL；WBC≥3*109/L，ANC≥1.5*109/L，PLT≥75*109/L
9. Men or women of childbearing age in the experiment are willing to take contraceptive measures
10. Estimated survival period for 3 months or more

Exclusion Criteria:

1. The palliative chemotherapy ever use docetaxel and pemetrexed
2. small cell lung cancer non small cell hybrid
3. Women during pregnancy or lactation
4. In the past the anti-tumor treatment of any outstanding ease of > CTCAE 2 levels of toxicity
5. Ccr<30 ml/min (calculated by Cockcroft-Gault formula)
6. hepatic insufficiency： Tbil> 1.5×ULN ALT and AST > 2.5×ULN (Patients with liver metastasis>5×ULN) Alkaline phosphatase>2.5 ×ULN(Patients with liver metastasis>5×ULN)
7. Severe symptomatic heart disease
8. Symptomatic brain metastases
9. In the last 5 years have been or are suffering from other histological types of malignant tumor
10. There are serious or uncontrolled systemic diseases
11. During the study period planned radiotherapy on target lesion
12. During the study period, plans to use other antineoplastic therapy
13. Clinical study on treatment of 30 days beginning period prior to participate in any study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Overall Officials: Chang J hua, PD, Principal Investigator — Fudan University
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China